CLINICAL TRIAL: NCT02633319
Title: Malezi ne Kilimo Bora (Good Parenting and Farming) - Skilful Parenting and Agribusiness Child Abuse Prevention Study (SPACAPS)
Brief Title: Malezi Na Kilimo Bora - Skilful Parenting and Agribusiness Child Abuse Prevention Study
Acronym: SPACAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Tanzanian National Institute of Medical Research (Unknown); University of Glasgow (Other); Investing in Children and Our Societies (Unknown); UBS Optimus Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: SSD/CUREC1A/14-SSH_C2_15_023
Record Dates: First submitted 2015-11-02; First posted 2015-12-17 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Child Abuse; Parenting
Keywords: Parenting; Child maltreatment; Economic strengthening; Early childhood development; Cluster randomized controlled trial; Pilot evaluation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Parenting Training (Experimental): Skilful Parenting: 12-week group-based parent intervention delivered by Investing in Children and Our Societies to caregivers who are members of farmer groups in participating villages.
  Interventions: Behavioral: Skilful Parenting
- Agricultural Training (Experimental): Agrics: Initial 3-month agricultural training intervention with ongoing support afterwards.
  Interventions: Other: Agrics
- Parenting and Agricultural Training (Experimental): Village farmer groups receiving both Skilful Parenting and Agrics interventions.
  Interventions: Behavioral: Skilful Parenting; Other: Agrics
- Control (No Intervention): 6-month wait-list control group

INTERVENTIONS:
Behavioral: Skilful Parenting — Skilful Parenting is a 2-week group-based parenting intervention delivered by Investing in Children and Our Societies to caregivers who are members of farmer groups in participating villages. It reinforces positive parenting practices, empowering parents to address the challenges that they face in bringing up their children. The intervention helps create parent peer groups to share ideas, support, information, and resources in the community. The intervention involves weekly sessions with farmer groups, awareness raising amongst local authorities and communities, and the establishment of parent peer groups. Topics consist of the following issues related to parenting: roles and responsibilities; family relations; communication; values; positive discipline; child protection; and family budgeting.
  Arms: Parenting Training; Parenting and Agricultural Training
Other: Agrics — Agrics provides smallholder farmers, organized in farmer groups, with access to farm inputs on a credit basis, and agricultural extension and advisory services to improve farming techniques and improve market connections. These services include an intensive intervention during planting season and then ongoing support after the initial 3-month intervention.
  Arms: Agricultural Training; Parenting and Agricultural Training

SUMMARY:
The Malezi ne Kilimo Bora ("Good Parenting and Farming" in Kiswahili) Skilful Parenting and Agribusiness Child Abuse Prevention Study is a collaboration between the University of Oxford, University of Glasgow, and the Tanzania National Medical Research Institute (NIMR). It is pilot cluster randomised controlled trial (cRCT) of a community-based intervention implemented by Investing in Children and Our Societies (ICS), an international non-governmental organization (NGO) with extensive experience operating in rural Tanzania. The overall focus of the project is to evaluate ICS's agribusiness and skilful parenting programmes' impact on the prevention of child maltreatment and improvement of child and family psychosocial and economic wellbeing (n = 8 villages, n = 16 farmer groups, n = 240 families).

DETAILED DESCRIPTION:
Background on Child Maltreatment in Tanzania

Child maltreatment and other childhood adversities often occur in many low- and middle-income countries at rates that are higher than in high-income countries - rates that often exceed 50%. In Tanzania, a national survey examining violence against children (VAC) found that almost 73.5% of females and 71.7% of males between the ages of 13 and 24 had experienced physical violence by prior to the age of 18. Furthermore, 23.6% of females and 27.5% of males had experienced emotional violence by an adult during childhood, and 27.9% of females and 13.4% of males had experienced some form of sexual violence before the age of 18 years. In addition, the survey identified an overlap among physical, emotional, and sexual violence against children. Approximately 80% of respondents who experienced sexual violence also experienced physical violence as a child, and nearly all children who experienced physical violence also experienced emotional violence. The VAC study also found that parents and other adult relatives are the most commonly reported perpetrators of physical and emotional violence against children, with corporal punishment considered a social norm.

Recent advances in neuroscience, genomics, developmental psychology, epidemiology, and economics have shed light on the long-term and far-reaching consequences of childhood adversities, many of which, like child maltreatment, are directly related to poor parenting. These consequences include serious physical and mental health problems later in life, as well as difficulties in school, jobs, and relationships. Child maltreatment can have substantial intergenerational effects in which some parents who experienced maltreatment during childhood are more vulnerable to the risk of maltreating their own children. Child maltreatment is also a risk factor for later intimate partner violence, increased risk of HIV-infection, and transactional sex amongst AIDS-affected youth. Furthermore, not only is child maltreatment a serious public health and human rights issue, but it comes at an economic cost due to expenses relating to the treatment of victims' health problems, criminal justice and welfare costs, and lower economic productivity.

The risks factors of child maltreatment can be best understood using an ecological framework. A recent review of 23 quantitative studies in Africa by Meinck et al identified a number of child, family, and social risk factors for child maltreatment. Child factors associated with increased likelihood of physical abuse included younger children, boys, children with disability or chronic illness, child behaviour problems, and school non-attendance and poor performance. Family-level factors include caregiver chronic illness, HIV/AIDS, caregiver mental health problems, caregiver disability, domestic violence, substance abuse, poor family functioning, and inconsistent parenting. Finally, household poverty and low socioeconomic status was found to be a major factor for increased risk of child abuse, as well as indirectly through increased family stress and reduced parental involvement.

Parenting Programmes to Prevent Child Maltreatment

Parenting programmes have shown particular promise in preventing child maltreatment and other childhood adversities and averting many of the life-long negative consequences for children and society. A recent meta-analysis reported that parenting programs successfully reduced substantiated and self-reported child maltreatment reports and reduced the potential for child maltreatment, both in high and middle-income countries. Often group-based, these programmes typically aim to strengthen caregiver-child relationships through play and praise, and to help parents to manage children's behaviour through effective, age-appropriate, positive discipline strategies. However, almost all the evidence for their effectiveness comes from high-income countries and they often cost many thousands of dollars per family served. They are thus prohibitively expensive for most governments and NGOs in low- and middle-income countries. Furthermore, their license-holders have been reluctant to implement them in such settings due to what they perceive as lack of the requisite infrastructure and trained personnel. In sum, there are currently no parenting programmes that are both evidence-based and affordable for low- and middle-income countries (LMIC), where the need is the greatest.

Economic Strengthening Programmes

Household poverty has also been identified as a risk factor for parental psychological distress and depression as well as physical and emotional child abuse. Consequently, in addition to improving parenting behaviour, in order to reduce the risk of child maltreatment, it may be necessary to address issues of poverty through economic strengthening programmes. These programmes include micro-financing, conditional and unconditional cash transfers, and agricultural interventions that provide skills training, credit loans, access to markets. However, there is still little empirical evidence on the benefits of an integrated approach of economic strengthening and parenting interventions. It may be sufficient to provide parent management training alone as a key mechanism of change in improving parent-child relationships and reducing the risk of child maltreatment. For instance, a recent meta-analysis by Leijten et al found that parenting programs were equally effective for socioeconomically disadvantaged families in comparison to non-disadvantaged families. On the other hand, some evidence suggests that families require additional support that addresses other social risk factors including poverty and material hardship. Furthermore, economic strengthening programs may in fact harm children if not combined with adequate child protection. Other research in East Africa indicates linkages between economic strengthening programs and child wellbeing, as well as the importance of integrating such interventions with psychosocial support. Nevertheless, more research is needed to understand the role of economic strengthening programs and parent management training in reducing on the risk of child maltreatment, as well as the utility of using a combined approach.

Study Aims and Design

This study aims to contribute to the literature on the prevention and reduction of child maltreatment in northern Tanzania. It will evaluate ICS's community-based intervention model that combines Agribusiness and Skilful Parenting training using a pilot cluster randomized controlled trial design (cRCT) in order to test intervention feasibility, acceptability, and preliminary efficacy. It will enable us to conduct both a process and rigorous outcome evaluation using a mixed-methods approach with qualitative focus groups and in-depth interviews combined with quantitative implementation data and self-report questionnaires.

This pilot cRCT will randomly allocate 8 villages (16 farmer groups, 2 farmer groups per village, 240 families, 20 families per farmer group) into the following four allocation groups (2 villages per allocation group):

1. Agribusiness only
2. Skilful Parenting only
3. Agribusiness plus Skilful Parenting
4. One-year wait-list control

For villages allocated to Agribusiness only, Skilful Parenting only, and/or the wait-list control group, participating farmer groups and families will have the opportunity to participate in the other intervention components after the final follow-up data assessment (1-year after baseline) provided that analysis of the results do not indicate any harmful effects.

This study will examine preliminary intervention effects comparing intervention arms with the wait-list control group as well as among active arms (Proschan, 1999). Although our focus will be on the effect of economic strengthening combined with parenting programs on reducing the risk of child maltreatment and improve child wellbeing, the investigators will also be examining the potential benefits of Skilful Parenting or Agribusiness programs delivered separately in comparison to controls.

This study will qualitatively and quantitatively examine intervention effects on parent-child interaction and child behaviour across the developmental spectrum. This includes (1) parents' report on interactions with a selected child between the ages of 3 to 17, (2) child report on parent-child interaction, child mental health, and child behaviour for families with children aged 10 to 16, and (3) early childhood development assessments in families with children aged 0 to 3. The investigators will also examine the feasibility (acceptability, implementation, and participation) of the Agribusiness and Skilful Parenting interventions.

Quantitative data collection will occur at 3 stages: baseline, immediate post-test, and 1-year follow-up from baseline. The investigators will use descriptive and psychometric scales to measure family socioeconomic status, parent-child interaction (including child maltreatment or harsh parenting), parent mental health, child depression and behaviour, early child development and stimulation, and child biometric data. Quantitative data collection will include parent report assessments for families with children aged 3 to 17, child report assessments for families with children aged 10 to 16, and early childhood development assessments for families with children aged 0 to 3. As a result, each participating family will have a maximum of 3 assessments per data collection stage.

Qualitative data will be collected from multiple sources using focus groups and in-depth interviews to strengthen the reliability of results: participating parents and co-parents, children, and facilitators. Focus groups (n=4) with participating families in the intervention arms will occur in local community centers at immediate post-test. In-depth interviews will take place at participants' homes with a targeted selection of participating parents, co-parents, and children (aged 10-16) at immediate post-test. In addition, focus groups will be conducted with program facilitators (n=8) at immediate post-test. Additional data will be collected from participants who drop out of the programme or have low attendance rates to examine barriers to participation.

Quantitative process data will be collected using trained staff responsible for monitoring programme facilitators. Weekly facilitator fidelity checklists will be administered after each session of Skillful Parenting. Research staff will also collect data on participant enrolment, participation, and engagement using attendance registers and client satisfaction surveys administered the end of program completion. This will allow us to quantitatively examine predictors of programme enrolment, participation, and dropout as well as potential risk factors for withdrawal from the intervention.

ELIGIBILITY:
Inclusion criteria for villages (n = 8):

1. Situated within 1 hour driving distance from Shinyanga, Tanzania
2. Provide community consent via community local leader and approval from local authorities
3. Contain registered farmer groups

Inclusion criteria for participating farmer groups (n = 16, 2 per village):

1. Situated within participating village
2. Registered with Tanzanian Ministry of Agriculture within the previous 3 years
3. Registered to participate in ICS's Agribusiness and Skilful Parenting programme
4. Provide consent via farmer group leader

Inclusion criteria for adults caregivers (n = 240, 30 per village):

1. Age 18 or older
2. Serves as the primary caregiver of a child in the household between the ages of 3 and 17
3. Lives in the house at least 4 nights per week.
4. Is a registered member of the included agricultural farmer group
5. Provides consent to participate in the full study

Exclusion criteria for adult participants:

1. Any adult exhibiting severe mental health problems or acute mental disabilities.
2. Any adult that has been referred to social services or child protection services during the course of baseline data collection as a result of reported or observed indications of significant potential psychological harm towards a child.

Inclusion criteria for child respondents (n = 240, 30 per village):

1. Age 10 to 17 years at initial assessment
2. Lives in the house at least 4 nights per week
3. Must have an adult primary caregiver who lives in the household, who provides consent, and who participates in the study
4. Provides assent to participate in the full study

Exclusion criteria for child respondents:

1. Any child who is either experiencing severe mental health problems, has acute developmental disabilities,
2. If the child participant has been referred to social services during baseline data collection due to reported or observed indications of significant harm.

Inclusion criteria for observed children (n = 240, 30 per village):

1. Age 0 to 3 years at initial assessment
2. Lives in the house at least 4 nights per week
3. Must have an adult primary caregiver who lives in the household, who provides consent, and who participates in the study

Inclusion criteria for adult ICS programme facilitators:

1. Age 18 or older
2. Is registered as a facilitator of ICS's Agribusiness or Skilful Parenting programme
3. Provides consent to participate in the full study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Child Abuse - Parent Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Child abuse will be measured using adapted versions of the ISPCAN Child Abuse Screening Tool-Parent version (ICAST-P), a multi-national and consensus-based survey instrument measuring the incidence and prevalence of child abuse and neglect. This 19-item scale ICAST-P was validated in 6 LMIC and 7 languages (α = 0.77-0.88) and measures four types of abuse: physical, emotional and sexual abuse, as well as neglect. In this study, the response code was adapted to a frequency scale from 0 to more than 8 times as certain behaviour occurred in the past month. In this study, incidence child maltreatment will be scored as dichotomous variables for physical, verbal, and sexual abuse, as well as an overall indication of previous child abuse (0 = no abuse; 1 = previous abuse). The investigators will also assess frequency of overall abuse by summing all of the subscales as well as for each individual subscale.
Change in Child Abuse - Child Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Child report of child abuse will be measured using adapted versions of the ISPCAN Child Abuse Screening Tool-Child version (ICAST-C), a multi-national and consensus-based survey instrument measuring the incidence and prevalence of child abuse and neglect. This 32-item scale ICAST-C was validated in 6 LMIC and 7 languages (α = 0.77-0.88) and measures four types of abuse: physical, emotional and sexual abuse, as well as neglect. In this study, the response code was adapted to a frequency scale from 0 to more than 8 times as certain behaviour occurred in the past month. In this study, incidence child maltreatment will be scored as dichotomous variables for physical, verbal, and sexual abuse, as well as an overall indication of previous child abuse (0 = no abuse; 1 = previous abuse). The investigators will also assess frequency of overall abuse by summing all of the subscales as well as for each individual subscale.
Change in Parenting Behaviour - Adult Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Parent-child interaction, will be measured using the Alabama Parenting Questionnaire (APQ) - Adult Report (37 items). The APQ contains five subscales assessing Positive Parenting (8 items), Parent Involvement (8 items), Inconsistent Discipline (11 items), Poor Supervision (10 items). The APQ has been shown to have moderate to strong internal reliability for both parent and child reports (Cronbach's α = 0.50 to 0.89). It has been used widely including in LMIC such as South Africa and Mexico. Caregivers report on the frequency of parenting behaviour based on a 4-point Likert scale (0 = never; 3 = Often, more than 5 times). Items are summed to create total frequency score (range 0 to 81) as well as for each subscale.
Change in Parenting Behaviour - Child Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Parent-child interaction, will be measured using the Alabama Parenting Questionnaire - Child Report (42 items). The APQ contains five subscales assessing Positive Parenting (8 items), Parent Involvement (8 items), Inconsistent Discipline (11 items), Poor Supervision (10 items), and Harsh Discipline (5 items). The APQ has been shown to have moderate to strong internal reliability for both parent and child reports (Cronbach's α = 0.50 to 0.89). It has been used widely including in LMIC such as South Africa and Mexico. Children report on the frequency of parenting behaviour based on a 4-point Likert scale (0 = never; 3 = Often, more than 5 times). Items are summed to create total frequency score (range 0 to 126) as well as for each subscale.

SECONDARY OUTCOMES:
Change in Parental Attitudes to Punishment | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  This study asked one question from the UNICEF Multiple Indicator Cluster Survey regarding parental attitudes to physical discipline based on a 5-point Likert scale of 0 to 4: "In order to bring up, raise up, or educate a child properly, the child needs to be physically punished." Caregivers report whether they disagree or agree with the statement (0 = disagree strongly; 4 = agree strongly).
Change in Parenting Stress - Adult Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Parenting stress will be assessed using the Parental Stress Scale (PSS; 18 items). PSS has been widely used to measure parenting stress, including in LMIC, such as Pakistan and China. The scale has also been used with non-parent caregivers such as grandparents. Caregivers report current positive attitudes (n = 8, e.g., "I feel close to my child") and negative attitudes (n = 10, e.g., "I feel overwhelmed by the responsibility of being a parent") related to parenting stress based on a five-point Likert scale (0 = strongly disagree; 4 = strongly agree). Positive items are reversed and then all items are summed to create a total parenting stress score (range 0 to 90).
Change in Caregiver Depression - Adult Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  The Centre for Epidemiological Studies Depression Scale (CES-D) (20 items) has been widely used throughout LMIC to assess self-report screening of adult depression. This was used in previous studies in sub-Saharan Africa of caregivers with strong reliability (α = .91). Caregivers report on the frequency of depressive symptoms in the previous week (0 to 7 times, e.g., "I thought my life was a failure"). Items are summed to create an overall depression score.
Change Child Behaviour - Adult Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Strengths and Difficulties Questionnaire has been used previously in Tanzania and has officially been translated into Kiswahili. It examines prosocial behaviour, conduct problems, hyperactivity-inactivity, peer problems, and emotional problems. The investigators also added a 5-item subscale to assess local cultural norms of child behaviour regarding respectability, or Hashima (e.g., "My child's behaviour brings embarrassment to my family"). Items are summed for each subscale (range 0 to 10). Behaviour problem subscales are also summed to create a total child behaviour problems score (0 to 50).
Change Child Behaviour - Child Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Strengths and Difficulties Questionnaire has been used previously in Tanzania and has officially been translated into Kiswahili. It examines prosocial behaviour, conduct problems, hyperactivity-inactivity, peer problems, and emotional problems. The investigators also added a 5-item subscale to assess local cultural norms of child behaviour regarding respectability, or Hashima (e.g., "My child's behaviour brings embarrassment to my family"). Items are summed for each subscale (range 0 to 10). Behaviour problem subscales are also summed to create a total child behaviour problems score (0 to 50).
Change in Intimate partner Violence - Adult Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  The Revised Conflict Tactics Scale Short Form (CTS2S; 10 items) measures exposure to intimate partner physical and psychological violence (IPV). Assessments use adult self-report on the frequency of negotiation, physical assault, psychological aggression, sexual coercion, and physical injury. Answers are coded on a 5-point Likert scale of 0 to 4 (0 = never happened; 4 = more than 3 times in the past month). The CTS2S will determine an overall indication of IPV on a level of severity (sum of items) and prevalence (dichotomous variable indicating experience of conflict or not) as well as for each subscale. The CTS2S has been used extensively in studies on IPV in sub-Saharan Africa. The original validation study showed strong internal consistency (α = .89).
Change in Child Labor - Adult Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Adult report of child involvement in labour will be measured using items from the UNICEF MICS Household Survey. This 6-item questionnaire asks caregivers whether their child was involved in farm work, running or helping to run a business, production of goods for sales, collection of firewood, or other household activities. It also assesses the amount of hours per week that the child is involved in each household task.
Change in Household Hunger - Adult Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Relative poverty will be assessed using 3 items from the Hunger Scale Questionnaire. These items examine food shortage and hunger in the household. Parents respond positively or negatively regarding the occurrence of hunger during the past 30 days and whether it occurred more than 5 times (e.g., "the household has run out of money to by food"). The scale produces scores for single occurrence and intensity of hunger.
Change in Agricultural Assets - Adult Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  In order to assess the impact of agribusiness training, household agricultural assets will be measured using 8 items from the UNICEF MICS Household Survey. Caregivers will be asked if the household owns land for farming and, if so, how many acres (individually, not collectively). They will also be asked which animals they own and how many (e.g., cattle).
Change in Household Assets - Adult Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Household assets will be assessed using items from the Economic Asset Index (9-items). The Economic Asset Index (EAI) measures relative household poverty based on methodology used in the Demographic Health Survey (DHS). This measurement has been used in over 55 countries, including Tanzania, and by the World Bank to asses relative poverty from a variety of factors. Instead of directly measuring poverty by income, the EAI examines adult reports of household ownership of consumer goods (cell phone, radio, car, etc.) and access to utilities and running water.
Change in Early Childhood Home Environment - Observed and Adult Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Observed early childhood home environment will be assessed using the Home Observation for Measurement of the Environment (HOME) assessment tool for infants and toddlers aged 0 to 3 years (44 items). It combines interview and observational items to assess the quality of family environment and engagement in child rearing. The scale includes 6 subscales: responsiveness (11 items), acceptance (7 items), organisation (6 items), play/learning materials (9 items), involvement (6 items), and variety of experience (5 items). The investigators eliminated one item on whether the family has a pet since it was considered culturally irrelevant. Double negative items on the Acceptance subscale were reversed to simplify the constructs. Assessors record whether the parent either reports the behaviour occurring or the behaviour is observed during the interview (0 = no; 1 = yes). Items are summed on each subscale as well as for an overall score on home environment stimulation and responsiveness.
Change in Child Development - Adult Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Child development will be assessed using the parent-report version of the Ages and Stages Questionnaire Version 3 (ASQ-3). This screening tool measures infant and toddler development from 2 months to 60 months (5 years) of age according to the following developmental domains: communication, gross motor, fine motor, problem-solving, and personal social skills. Each domain has 6 items (30 items in total). Distinct questionnaires are administered according to the child's age in 2-month intervals rounded to the nearest interval. The ASQ-3 is administered via caregiver self-report based on "Yes," "Sometime," or "Not Yet" for each developmental milestone. In addition, if the caregiver is not sure of a specific item, they are given the opportunity to perform the task with their infant or toddler. The entire assessment takes approximately 20 minutes. Items for each subscale are summed to create total scores as well as an overall indication of child development.
Change in Infant/Toddler Weight | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Child weight will be determined using a 25 kg Salter hanging scale (Weighing equipment, High Holborn, London, United Kingdom) with the child in light clothes and no shoes. A standard beam balance (SECA) will be used in weighing the young infants. The readings will be recorded to the nearest 0.1kg. Calibration of weighing scale to zero will be performed every day during the assessment period. A known 1kg weight will be used to standardize the scales every day for accuracy and consistency.
Change in Infant/Toddler Height | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Child height will be measured using a length board. Children will be placed lying shoeless in the supine position on the board with their heads placed at 900 to the fixed head piece. Research assistants will straighten the legs of the child at the knees and ensured that feet were at right angle to the sliding foot piece, which will be brought into contact to the child's heels. Child length will be recorded to the nearest 0.1 centimeters.
Change in Household Hunger - Child Report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Child report on relative poverty will be assessed using 3 items from the Hunger Scale Questionnaire. These items examine food shortage and hunger in the household. Children will be asked to respond positively or negatively regarding the occurrence of hunger during the past 30 days and whether it occurred more than 5 times (e.g., "the household has run out of money to by food"). The scale produces scores for single occurrence and intensity of hunger.
Change in Child food consumption - Child report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  This study will assess consumption via child report on average meals consumed per day in the past week based on items from the UNICEF MICS Household Survey (e.g., "how many meals did the participant consumer per day").
Change in Child labour - Child report | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Child involvement in labour will be measured using items from the UNICEF MICS Household Survey. This 6-item questionnaire asks children whether they were involved in household chores, farm work, running or helping to run a business, production of goods for sales, collection of firewood, or other household activities in the past week. It also assesses the amount of hours per week that the child is involved in each household task.
Change in Child Attitudes to Punishment | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  This study asked one question from the UNICEF Multiple Indicator Cluster Survey regarding parental attitudes to physical discipline based on a 5-point Likert scale of 0 to 4: "In order to bring up, raise up, or educate a child properly, the child needs to be physically punished." Children report whether they disagree or agree with the statement (0 = disagree strongly; 4 = agree strongly).
Change in Child Depression | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Child depressive symptoms will be measured using the 10-item Child Depression Inventory (CDI) short form. This was used previously with vulnerable children in sub-Saharan Africa including a recent cross-cultural adaptation in in Kiswahili in rural Tanzania. Each item is scored on a three-point scale (0 absent; 1 moderate; 2 severe) according to symptom severity with a total possible score ranging from 0 to 20. The Tanzanian study showed acceptable reliability (α = .66).
Change in Child Sexual Behavior | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Sexual behaviour Child sexual behaviour will be measured using 15 items from the South African National Survey of HIV and risk behavior amongst young South Africans. This study will measure sexual debut, concurrent sexual partners, sexual activity under the influence of alcohol and under the influence of drugs, and pregnancy. These items have been used in previous studies on youth in sub-Saharan Africa. In the current study, the time period was adapted to the past month to be appropriate for the present RCT research project.
Change in Child Alcohol Use | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Child use of alcohol will be assessed by measuring alcohol consumption during the past month (1 item). Due to the sensitive nature of these items, additional items dealing with other activities to reduce stress have been included in this section to encourage accuracy (2 items; e.g., "In the past month, did the particpant play sports or dance with friends to relax?").
Change in Adult Alcohol Use | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Parental dependency on alcohol will be assessed by measuring alcohol consumption during the past month (1 item). Dependency is based on 3 or more drinks per day for female participants and 5 or more per day for male participants. Due to the sensitive nature of these items, additional items dealing with other activities to reduce stress have been included in this section to encourage accuracy (3 items; e.g., "In the past month, has the participant been for a walk or done some other exercise to help the participant relax?").

OTHER OUTCOMES:
Basic Caregiver and Child Demographic Information | Baseline
  Basic caregiver and child demographic information will be asked using items from the UNICEF Multiple Indicators Cluster Survey (MICS) Household Survey. It assesses caregiver/child age, gender, marital status, employment status, education level, basic literacy, child's relationship to caregiver, presence of child's biological parents (including reasons for absence), and other household members' age, gender and relationship to caregiver. It also assesses other household socio-demographic characteristics including household structure, family employment, and whether or not the family receives any governmental grant support.
Change in Caregiver General Health | Baseline; 6-Months Follow-Up; 12-Months Follow-Up
  Caregiver general health will be assessed using 3 items from the Medical Outcomes Study (MOS) Short Form-12 Health Survey (SF-12). This scale is an adapted version of the MOS SF-34 Health Survey to examine physical and mental health. Items include difficulty in moderate daily activities, such as moving boxes, shopping, or carrying a child. Response options are based on a 3-point Likert-like scale (1 = yes, limited a lot; 3 = no, not limited at all). An additional item requires respondents to assess their overall health on a 5-point Likert scale (1 = excellent; 5 = poor).
Caregiver/Child Disability | Baseline
  Caregiver and child disability will be assessed using the census questions (4 items) on disability endorsed by the Washington Group. These questions rely on self-report of difficulty the caregiver or child may experience in seeing, hearing, walking or climbing steps, remembering, washing him/herself, and communicating in his/her usual language. Response options have been simplified to "yes" or "no" for each item. Two additional items asks respondents whether they or their child has a disability. If they respond "yes", they are asked to specify which type of disability.
Parental History of Child Maltreatment | Baseline
  Parental history of child maltreatment in their families of origin will be measured using an adapted version of the ISPCAN Child Abuse Screening Tools Retrospective version (ICAST-R, 10 items). This scale utilises parent self-report of experiences during their own childhood (under 18 years old) to assesses the history of incidence of physical maltreatment, verbal abuse, and sexual abuse. In this study, incidence of past history of child maltreatment will be scored as dichotomous variables for physical, verbal, and sexual abuse, as well as an overall indication of previous child abuse (0 = no abuse; 1 = previous abuse).
Obstacles to Engagement Scale | Baseline
  Adult report of barriers to program participation and engagement will be measured using the Obstacles to Engagement Scale. This 14-itme scale has four subscales: family obstacles (4 items); relevance of parenting programmes (4 items); suitability of group-based programmes (4 items); and barriers due to time commitments (2 items). Participants rate each item on a 7-point sliding Likert scale ranging from "Strongly disagree" to "Strongly agree." Scores for each subscale are created as well as an overall barrier to engagement score by summing totals.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Gardner, DPhil, Principal Investigator — University of Oxford; Joyce Wamoyi, PhD, Principal Investigator — Tanzania National Institute of Medical Research
Locations (1):
- Tanzania National Institute of Medical Research, Mwanza, Tanzania

REFERENCES:
- [Derived] Lachman J, Wamoyi J, Spreckelsen T, Wight D, Maganga J, Gardner F. Combining parenting and economic strengthening programmes to reduce violence against children: a cluster randomised controlled trial with predominantly male caregivers in rural Tanzania. BMJ Glob Health. 2020 Jul;5(7):e002349. doi: 10.1136/bmjgh-2020-002349. PMID 32641291